CLINICAL TRIAL: NCT06186986
Title: Molecular Imaging of Zirconium-89-labeled Brentuximab as a Tool to Investigate Brentuximab Biodistribution in CD30-positive Lymphoma
Brief Title: CD30 Imaging in Diffuse Large B-cell Lymphoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Medical Center Groningen (Other)
Collaborators: Takeda (Industry)
Responsible Party: Principal Investigator, Marcel Nijland, Hematologist, University Medical Center Groningen
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: NL202100762
Record Dates: First submitted 2023-10-05; First posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Diffuse Large B-cell-lymphoma
MeSH Terms: conditions — Dendritic Cell Sarcoma, Interdigitating | interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Part 1 (Experimental): In Part 1 of this side study a minimum of 5 eligible patients will undergo 89Zr-brentuximab-PET scans at 3 different time points (1, 4 and 7 days after tracer injection) either without (2 patients) or with preceding administration of 10 mg (3 patients) or more (n patients) of unlabeled brentuximab.
  Interventions: Drug: Brentuximab vedotin
- Part 2 (Experimental): In Part 2 of this side study the optimized imaging schedule from Part 1 will be used to investigate biodistribution and tumor uptake of 89Zr-brentuximab in 15 patients and correlate imaging data to baseline sCD30 serum levels, CD30 IHC and CD30 Gene Expression Profiling (GEP).
  Interventions: Drug: Brentuximab vedotin

INTERVENTIONS:
Drug: Brentuximab vedotin — 5 Participants will receive unlabeled brentuximab and 20 participants will receive 89ZR-Brentuximab.
  Other Names: 89ZR-Brentuximab

SUMMARY:
The antibody drug conjugate (ADC) brentuximab vedotin (BV), targeting CD30, is currently registered for the treatment of previously untreated stage III-IV Hodgkin lymphoma (HL), relapsed Hodgkin lymphoma, relapsed systemic anaplastic large T-cell lymphoma (sALCL) and relapsed CD30 expressing cutaneous T-cell lymphoma, type mycosis fungoides (CTCL, MF) with overall response rates (ORR) up to 70%. BV has shown promising results in other CD30 expressing non-hodgkin lymphoma (NHL), including relapsed angio-immunoblastic T-cell lymphoma (AITL), peripheral T-cell lymphoma not otherwise specified (PTCL-NOS), post-transplant lymphoproliferative diseases (PTLD) and diffuse large B-cell lymphoma (DLBCL) with ORR rates of 50%, 40% and 45%, respectively. Despite expression of CD30 on tumor cells, no objective responses were observed in relapsed primary mediastinal B-cell lymphoma (PMBCL). Strikingly, thus far correlative studies have not found predictive markers in tissue or blood that are predictive for response to treatment. Since CD30 expression in tumor tissue is unrelated to treatment outcome, this suggests involvement of phenomena like tumor heterogeneity, drug uptake in the tumor micro-environment or very low CD30 expression below the immunohistochemistry (IHC) threshold. In this imaging study the biodistribution of brentuximab will be investigated by using Zirconium-89 (89Zr)-labeled brentuximab. 89Zr-brentuximab imaging will help to assess tumor uptake and pharmacokinetic (PK) and -dynamic properties of brentuximab in patients who are intended to be treated with BV, either in one of the registered indications (HL, CTCL and sALCL) or as part of the HOVON 136 trial for patients with DLBCL. The hypothesize is that the results of this imaging study might be used to facilitate the identification of patients that would benefit most from BV treatment

ELIGIBILITY:
Inclusion Criteria:

* All patients with histologically proven CD30-positive (i.e. > 1% cells) lymphomas who will be treated with BV, including:

  * HL
  * T-NHL
  * CTCL
  * DLBCL

    * Age ≥18 years
    * Signed written informed consent form (approved by the Institutional Review Board [IRB]/ Independent Ethics Committee [IEC]) obtained prior to any study specific screening procedures
    * Measurable disease: on CT scan at least 1 lesion/node with a long axis of > 1.5 cm and at least one positive lesion on 18F-FDG PET scan
    * World Health Organization (WHO) performance status 0-2 (see appendix A)
    * Adequate hepatic function: total bilirubin ≤ 1.5 times upper limit of normal (ULN) (unless due to lymphoma involvement of the liver or a known history of Gilbert's syndrome as defined by > 80% unconjugated bilirubin) and Alanine Aminotransferase (ALAT) / Aspartate Aminotransferase (ASAT) ≤ 3 times ULN (unless due to lymphoma involvement of the liver; in that case ALAT/ASAT may be elevated up to 5 times ULN)
    * Adequate renal function: GFR > 50 milliliter/ minute (ml/min) as estimated by the cockcroft & gault formula at rehydration:

Creatinine Clearance (CrCL) = (140-age [in years] x weight [kg] (x 0.85 for females) (0.815 x serum creatinine [μmol/L])

* Adequate bone marrow function: Absolute neutrophil count (ANC) ≥ 1.5 x 109/liter (L) and platelet count ≥100 x 109/L, unless caused by diffuse bone marrow infiltration by lymphoma
* Hemoglobin must be ≥ 8 g/dL (5.0 mmol/L), transfusion is allowed
* Life expectancy of >3 months with treatment
* Negative pregnancy test at study entry, if applicable

Exclusion Criteria:

* Prior allergic reaction or known hypersensitivity to immunoglobulins, recombinant proteins, murine proteins, or to any excipient contained in the dug formulation of BV.

  * Peripheral sensory or motor neuropathy grade ≥ 2
  * Patients with a serious psychiatric disorder that could, in the investigator's opinion, potentially interfere with the completion of treatment according to protocol
  * Patients who have any severe and/or uncontrolled medical condition or other conditions that could affect their participation in the study
  * Any psychological, familial, sociological and geographical condition potentially hampering compliance with the study protocol and follow-up schedule
  * Claustrophobia to the extent that PET-CT is impossible
  * Pregnant or lactating women. Documentation of a negative pregnancy test must be available for pre-menopausal women with intact reproductive organs and for women less than two years after menopause

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
An optimized 89Zr-brentuximab imaging protocol for visualisation of CD30 distribution by PET-scan | 2 years
  89Zr-brentuximab imaging protocol, including the dose of brentuximab (mg), the dose of 89Zr-brentuximab (mg) and the time (day) of PET-scanning after 89Zr-brentuximab administration
Safety profile of the 89Zr-brentuximab tracer | 2 years
  AE related to imaging protocol with the 89Zr-brentuximab tracer
Relation 89Zr-brentuximab biodistribution and CD30 expression | 2 years
  Relation between 89Zr-brentuximab tracer uptake and CD30 protein expression

SECONDARY OUTCOMES:
Relation between 89Zr-brentuximab uptake and response to therapy | 2 years
  The extent of heterogeneity in 89Zr-brentuximab uptake and the potential correlation with response to therapy (as determined via 18F-FDG PET/CT scan per the International Working Group criteria (1,2).

CONTACTS AND LOCATIONS:
Overall Officials: Marcel Nijland, MD, Principal Investigator — UMCGoningen

IPD SHARING:
Plan to Share IPD: No
all IPD that underlie results in a publication